CLINICAL TRIAL: NCT05698589
Title: Compassion Focused Therapy (CFT) for the Reduction of the Internalized Stigma of Mental Disorders: a Multi-center, Prospective, Randomized, Controlled Study
Brief Title: COMpassion for Psychiatric Disorders And Self-Stigma
Acronym: COMPASS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8566
Record Dates: First submitted 2022-12-09; First posted 2023-01-26 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Bipolar Disorder; Schizophrenia; Depression; Borderline Personality Disorder; Autism Spectrum Disorder
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia; Depression; Borderline Personality Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Compassion Focused Therapy (Experimental)
  Interventions: Behavioral: Compassion Focused Therapy
- Ending Self Stigma (Active Comparator)
  Interventions: Behavioral: Ending Self Stigma
- Treatment As Usual (No Intervention)

INTERVENTIONS:
Behavioral: Compassion Focused Therapy — CFT is an experiential therapy. As such, in addition to psychoeducation components (e.g.: compassion from an evolutionary and neuroscientific perspective, the tricky brain problem, emotion regulation systems) and explicit learning of emotion regulation skills (in particular, shame), experiential exercises are provided in-sessions (e.g. : chair work, role plays, guided mental imagery, …) and between sessions practices will be provided with video guides, made available for the participants online (e.g. : soothing rhythm breathing, safe place imagery, compassionate self-imagery, …). The overall aim of the CFT program is to help participants shift from a hostile and critical self-to-self relationship to a more compassionate relationship to self.
  Arms: Compassion Focused Therapy
Behavioral: Ending Self Stigma — Psychoeducation sessions cover topics such as the path from public stigma to self-stigma and modifying self-stigmatizing thoughts. Participants will be encouraged to do home practices (e.g. writing about the pros and cons of self-stigmatizing thoughts) between sessions. The overall aim of the ESS program is to help participants address self-stigma with concrete tools to increase their self-esteem and achieve their goals
  Arms: Ending Self Stigma

SUMMARY:
People with mental disorders face frequent stigmatizing attitudes and behaviors from others . In response to this, they tend to isolate themselves, with the risk of impeding care and the process of recovery and integration into society . Stigmatization can also be assimilated by patients themselves - i.e. self-stigma. Self-stigma is involved in diminished coping skills that lead to social avoidance and difficulties in adhering to care . Reducing self-stigma and its emotional corollary, shame, is thus crucial to attenuate the disability associated with mental illness. Shame is inherent to self-stigma and leads to difficulties in adhering to care as well as greater severity of clinical presentations . Compassion Focused Therapy (CFT) is a third wave cognitive behavioral therapy that targets shame reduction and hostile self-to-self relationship and allows for symptom improvement while increasing self-compassion, a major resilience factor . Although shame is a prominent part of the concept of self-stigma, the efficacy of CFT has never been evaluated in individuals with high levels of self-stigma.

In this study, the investigators will evaluate the efficacy and acceptability of a group based CFT program on decreasing self-stigma, compared to treatment as usual (TAU) and a psychoeducation program whose efficacy has been assessed in a previous trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥18 years of age
2. Patient informed of the results of the preliminary medical examination
3. Patient affiliated to a social health insurance plan (beneficiary or beneficiary's family)
4. Patient with one or several diagnoses of chronic psychiatric disorder (schizophrenia, schizoaffective disorder, bipolar disorder, recurrent major depression, borderline personality disorder) or a neurodevelopmental disorder (autism spectrum disorder) treated as an outpatient or in a day hospital
5. CGI-Severity score<6 assessed by the psychiatrist (Berk et al., 2008) ISMI score indicating moderate to high self-stigma (>2.5; Lysaker et al., 2007)

   Exclusion criteria:
6. Patient in an exclusion period determined by a previous or ongoing study
7. Patient participating in an interventional study involving psychotherapy or an experimental drug
8. Patient in acute episode of their disorder according to the CGI Severity score
9. Patient in a medical emergency or immediate life-threatening situation
10. Patients with an intellectual disability (IQ<70) estimated via the fNART (Mackinnon & Mulligan, 2005)

12. Legal issues: care under constraint or patient deprived of freedom because of a judicial measure 13. Patient who does not speak and read French sufficiently

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Internalized Stigma of Mental Illness inventory (ISMI) | Day 0
  ISMI is : Internalized Stigma of Mental Illness Scale , The participant must select their response on a 4-point Likert scale ranging from strongly disagree (1) to strongly agree (4), hence the minimum and maximum score values are respectively 1 and 4. Higher scores mean worse outcome
Internalized Stigma of Mental Illness inventory (ISMI) | Month 1
  ISMI is : Internalized Stigma of Mental Illness Scale , The participant must select their response on a 4-point Likert scale ranging from strongly disagree (1) to strongly agree (4), hence the minimum and maximum score values are respectively 1 and 4. Higher scores mean worse outcome
Internalized Stigma of Mental Illness inventory (ISMI) | Month 2
  ISMI is : Internalized Stigma of Mental Illness Scale , The participant must select their response on a 4-point Likert scale ranging from strongly disagree (1) to strongly agree (4), hence the minimum and maximum score values are respectively 1 and 4. Higher scores mean worse outcome
Internalized Stigma of Mental Illness inventory (ISMI) | Month 3
  ISMI is : Internalized Stigma of Mental Illness Scale , The participant must select their response on a 4-point Likert scale ranging from strongly disagree (1) to strongly agree (4), hence the minimum and maximum score values are respectively 1 and 4. Higher scores mean worse outcome

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Pôle de Psychiatrie Adulte, Hôpital Charles Perrens, Bordeaux
  - Ch Le Vinatier, Bron
  - CHU de Clermont-Ferrand, Hôpital Gabriel Montpied, Service de Psychiatrie B, Clermont-Ferrand
  - Pôle Hospitalo-Universitaire de Psychiatrie d'adultes et d'addictologie du Grand Nancy, Centre Psychothérapique de Nancy, Laxou
  - CHU de Montpellier, Psychiatrie d'adultes, Hôpital la Colombière, Montpellier
  - Etablissement Public de Santé Mentale (EPSM) de la Marne, Site Pierre-Briquet, Unité de réhabilitation psychosociale, Reims
  - Service de Psychiatrie, Hôpital Civil, Hôpitaux Universitaires de Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Riebel M, Rohmer O, Charles E, Lefebvre F, Weibel S, Weiner L. Compassion-focused therapy (CFT) for the reduction of the self-stigma of mental disorders: the COMpassion for Psychiatric disorders, Autism and Self-Stigma (COMPASS) study protocol for a randomized controlled study. Trials. 2023 Jun 12;24(1):393. doi: 10.1186/s13063-023-07393-y. PMID 37309006